CLINICAL TRIAL: NCT00746369
Title: IMARA, Adapting SiHLE for Detained African American Adolescent Females
Acronym: IMARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00005355; 5UR6PS000679 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: HIV; Prevention; Adolescents; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention)
- Intervention (Experimental): IMARA HIV Prevention Intervention. Three individual sessions for incarcerated female teens.
  Interventions: Behavioral: IMARA HIV Prevention Intervention

INTERVENTIONS:
Behavioral: IMARA HIV Prevention Intervention — Three individual sessions- behavioral intervention for incarcerated female adolescents.
  Arms: Intervention

SUMMARY:
The IMARA Program will test the efficacy of a multi-session HIV Prevention program, adapted from an existing program(SiHLE), for incarcerated African American adolescent females.

DETAILED DESCRIPTION:
African American adolescent females in youth detention centers are at high risk for HIV infection. There are, however, no evidence-based interventions (EBI) for this vulnerable population. The aim of this project is to develop and test a culturally and gender-appropriate sexual health education program designed to promote HIV preventive sexual behaviors among African American adolescent females in youth detention centers. The study will be conducted in four stages: (1) adaptation of SiHLE intervention; (2) pilot adapted intervention; (3) revisions to adapted intervention, measures, and implementation; and (4) implementation and evaluation.

We will work closely with the Metro Regional Youth Detention Center (RYDC), in Atlanta, Georgia for all four stages of the project. The first stage, adaptation of SiHLE intervention, will be implemented using data collected from a prior study and with use of Community and Teen Advisory Boards (CAB and TAB). The pilot intervention will be completed with 20 participants from Metro RYDC and will test recruitment and retention strategies, the adapted intervention, and all measures. Revisions will be made based on findings from the pilot. For stage four, implementation and evaluation, we propose to recruit 350 unmarried African American adolescent females, 13-17 years of age, from Metro RYDC. While at the Metro RYDC, adolescents will be invited to participate in the proposed study. All adolescents will be required to have verbal informed parental/guardian consent and complete signed assent forms. Adolescents who are eligible and willing to participate in the project will complete an initial survey conducted on a computer(ACASI). The survey is designed to assess adolescents' sexual risk and preventive behaviors. After they complete the survey, adolescents will then be assigned, by chance alone, to receive either the adapted SiHLE intervention or the control condition. All adolescents will complete 3 individual sessions implemented by an African American health educator.

As we anticipate the participants will be released prior to the follow-up assessment, adolescents will come to a central community site to complete follow-up interviews at 3 and 6-months after completing their initial survey. We will also obtain a self-collected vaginal swab specimen to test for chlamydia and gonorrhea. We will compare the new adapted SiHLE intervention, IMARA, to the control condition in its ability to maintain or enhance adolescents' use of HIV prevention behaviors. If successful, the findings could have important implications for HIV prevention in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* African American
* Ages 13-17
* Sexually experienced
* Incarcerated at least 2 days and released to a non-restrictive setting
* Parent/guardian consent
* Assent

Exclusion Criteria:

* Married
* Pregnant

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proportion of condom protected vaginal sex acts over the last 90 days | 3 and 6 months post-randomization

SECONDARY OUTCOMES:
Incident infection of chlamydia or gonorrhea as confirmed by laboratory PCR testing | 3 and 6 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J. DiClemente, PhD, Principal Investigator — Emory University
Locations (1):
- Metro Regional Youth Detention Center, Atlanta, Georgia, United States

REFERENCES:
- [Background] Latham TP, Sales JM, Boyce LS, Renfro TL, Wingood GM, DiClemente RJ, Rose E. Application of ADAPT-ITT: adapting an evidence-based HIV prevention intervention for incarcerated African American adolescent females. Health Promot Pract. 2010 May;11(3 Suppl):53S-60S. doi: 10.1177/1524839910361433. PMID 20488969
- [Background] Latham TP, Sales JM, Renfro TL, Boyce LS, Rose E, Murray CC, Wingood GM, DiClemente RJ. Employing a teen advisory board to adapt an evidence-based HIV/STD intervention for incarcerated African-American adolescent women. Health Educ Res. 2012 Oct;27(5):895-903. doi: 10.1093/her/cyr003. Epub 2011 Mar 2. PMID 21368023